CLINICAL TRIAL: NCT01055925
Title: Clinical Comparative Trial of a Modified Polyurethane Dressing and Aquacel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik Bogenhausen (Other)
Purpose: Treatment
Other Study IDs: MPV-AQUACEL
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Reepithelialization of Skin Graft Donor Sites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MPV (Active Comparator)
  Interventions: Device: modified polyurethane film dressing (OpSite, Smith&Nephew, London, UK)
- Aquacel (Active Comparator)
  Interventions: Device: Aquacel® (ConvaTec, Skillman, NJ, USA), sodium carboxy-methylcellulose hydrocolloid polymer dressing

INTERVENTIONS:
Device: modified polyurethane film dressing (OpSite, Smith&Nephew, London, UK)
  Arms: MPV
Device: Aquacel® (ConvaTec, Skillman, NJ, USA), sodium carboxy-methylcellulose hydrocolloid polymer dressing
  Arms: Aquacel

SUMMARY:
The almost single disadvantage of conventional polyurethane film dressings, an uncontrolled leakage, is probably as often described as its numerous advantages for split-thickness skin graft (STSG) donor sites. This shortcoming can be overcome by perforating the polyurethane dressing (MPD), which permits a controlled leakage into a secondary absorbent dressing. The study was conducted to compare the MPD-system and Aquacel® (ConvaTec), a hydrofiber wound dressing, which also seems to fulfill all criteria of an ideal donor site dressing.

ELIGIBILITY:
Inclusion Criteria:

* skin graft donor site anterolateral thigh
* men and women > 18 years

Exclusion Criteria:

* informed consent missing
* repeated skin graft take or prior injury at the observed site
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* History of hypersensitivity to the investigational products

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
reepithelialization rate | 10th day postoperative

SECONDARY OUTCOMES:
pain, scar formation, complications (e.g. infection), costs | pain until and during dressing removal, scar formation 60 days following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Plastic, Reconstructive, Hand and Burn Surgery, Academic Hospital Munich Bogenhausen, Technical University Munich, Munich, Bavaria, Germany